CLINICAL TRIAL: NCT02935270
Title: Examining Measurement of Behavioral Neglect Post Stroke
Status: Completed | Type: Observational
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Michelle Woodbury, Post Doctoral Scholar, Medical University of South Carolina
Other Study IDs: PR00044531
Record Dates: First submitted 2016-10-12; First posted 2016-10-17 (Estimated); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Stroke; Hemispatial Neglect
Keywords: Stroke; Neglect; Rehabilitation
MeSH Terms: conditions — Stroke; Perceptual Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Stroke Survivors: Individuals who have experienced a unilateral hemispheric stroke

SUMMARY:
The purpose of this study is to examine measurement of unilateral neglect post stroke. Although a number of clinical assessments are used to measure neglect, it is unclear whether items from some of the most commonly used assessments are able to effectively and comprehensively measure neglect. This study will determine whether these assessments measure different aspects of neglect and whether items from various neglect assessments can be combined to more effectively measure neglect.

DETAILED DESCRIPTION:
Many individuals have difficulty attending to the affected side of their body or to the affected side of space after stroke (unilateral neglect). Although a number of clinical assessments are used to measure this inattention, it is unclear whether items from some of the most commonly used assessments are able to effectively and comprehensively measure inattention. Clinical assessments provide critical information to clinicians and researchers and are used to inform treatment and document patient progress. Therefore, it is important that investigators more closely examine these existing assessments.

Individuals who demonstrate impaired attention to the affected side after stroke also have greater motor impairment than individuals who do not have impaired attention, but investigators do not know how inattention affects reaching movements using the impaired arm. This study will examine various methods used to assess inattention to the affected side after stroke and also examine how inattention affects reaching movements of the impaired arm.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral hemispheric stroke
* 18 years or older

Exclusion Criteria:

* Severe aphasia
* Inability to follow 2-step directions
* Presence of other neurological disease that may impair vision or perception during performance of evaluation procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stroke survivors
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2016-01; Primary Completion 2020-02-21 (Actual); Study Completion 2020-02-21 (Actual)

PRIMARY OUTCOMES:
Catherine Bergego Scale | One-time assessment scheduled over 1-2 days
Behavioral Inattention Test | One-time assessment scheduled over 1-2 days
Naturalistic Action Test | One-time assessment scheduled over 1-2 days
Virtual Reality Lateralized Attention Test | One-time assessment scheduled over 1-2 days
Kinematic Assessment of Arm Movement | One-time assessment scheduled over 1-2 days

SECONDARY OUTCOMES:
Arm Use measured by Accelerometers | One-time assessment scheduled over 3 days
  Accelerometers will be issued on the first assessment day. Participants will wear accelerometers for 3 days.

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Woodbury, PhD, OTR/L, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Grattan ES, Woodbury ML. Do Neglect Assessments Detect Neglect Differently? Am J Occup Ther. 2017 May/Jun;71(3):7103190050p1-7103190050p9. doi: 10.5014/ajot.2017.025015. PMID 28422631